CLINICAL TRIAL: NCT03579160
Title: Efficacy and Safety of 0.25% Timolol Gel in Enhancing Full Thickness Skin Grafts Healing and Cosmetic Outcomes: A Randomized, Controlled Trial
Brief Title: Efficacy and Safety of 0.25% Timolol Gel in Enhancing Full Thickness Skin Grafts Healing and Cosmetic Outcomes
Acronym: FTSG
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the insufficient accrual rate and strategic reasons to focus our efforts on higher impact research projects.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Chrysalyne D Schmults, MD, MSCE, Director, Mohs and Dermatologic Surgery Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BWHMDSC003
Record Dates: First submitted 2018-06-07; First posted 2018-07-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Wound of Skin; Wound Heal; Surgical Wound; Full Thickness Skin Graft Healing
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: The protocol will begin post-surgery. Eligible subjects will be assigned by computer-based randomization to case (0.25% timolol gel) or control (standard of care [SOC]) group and treated as follows:
  Receiving site of FTSG/case group:
  1. During surgery: application of 0.25% timolol gel (2 drops per cm2) on wound bed before FTSG is placed
  2. During surgery: application of 0.25% timolol gel (2 drops per cm2) over FTSG after insetting of the graft
  3. After bolster removal (7 days): daily cleansing and daily 0.25% timolol (2 drops per cm2) application for 4 weeks
  Receiving site of FTSG/control group:
  1. FTSG surgery as per SOC
  2. After bolster removal (7 days): daily cleansing and daily Vaseline application for 4 weeks
Who Masked: Outcomes Assessor
Masking Description: Blinded physician will assess outcomes from pictures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 0.25% Timolol gel applied to full-thickness skin graft (Experimental): 1. During surgery: application of 0.25% timolol gel (2 drops per cm2) on wound bed before FTSG is placed
  2. During surgery: application of 0.25% timolol gel (2 drops per cm2) over FTSG after insetting of the graft
  3. After bolster removal (7 days): daily cleansing and daily 0.25% timolol (2 drops per cm2) application for 4 weeks
  Interventions: Drug: 0.25% timolol gel with full-thickness skin grafts
- Standard of Care dressings (Active Comparator): 1. FTSG surgery as per SOC
  2. After bolster removal (7 days): daily cleansing and daily Vaseline application for 4 weeks
  Interventions: Other: Vaseline dressing

INTERVENTIONS:
Drug: 0.25% timolol gel with full-thickness skin grafts — Timolol 0.25% gel will be applied to wound bed immediately after surgery before dressing is applied.
  Arms: 0.25% Timolol gel applied to full-thickness skin graft
Other: Vaseline dressing — Vaseline will be applied to wound bed immediately after surgery before dressing is applied.
  Arms: Standard of Care dressings

SUMMARY:
The use of topical beta-blockers, such as 0.25% timolol, in promoting wound healing is currently emerging in the academic literature. The investigators will enroll 82 patients who have their skin cancer surgically removed resulting in the need of a full-thickness skin graft. The objective of this randomized safety study is to determine the safety and efficacy of 0.25% timolol in promoting wound healing in full-thickness skin grafts compared to standard of care.

DETAILED DESCRIPTION:
The role of topical beta-blockers in promoting wound healing is currently emerging in the international literature. β2-Adrenergic receptors (B2AR) are the only subtype of beta-adrenoceptors expressed on skin. They can be found in secretory coil of apocrine glands, keratinocytes, fibroblasts and melanocytes. The distribution of these receptors provides insight on dermatological disorders that may be affected by β-blockers. Keratinocyte migration occurs by the facilitation of chemotaxis, the polarization of cells, and activation of extracellular signal-related kinases essential in the signaling of promigratory pathways. The B2AR activation inhibits keratinocyte migration by activating the serine/threonine phosphatase-2a, which downregulates phosphorylation of extracellular signal-related kinases necessary for migration. Therefore, B2AR antagonists prevent the phosphorylation of phosphatase-2a and have the downstream effect of extracellular signal-related kinase promotion, inducing a promigratory pathway in keratinocytes. Keratinocyte migration also occurs by galvanotaxis, a phenomenon in which cells migrate in response to electric stimuli. Keratinocytes can be stimulated to migrate with the formation of electrical poles and the application of electrical fields. The B2AR antagonists improve the ability of keratinocytes to respond to such migratory cues, whereas the B2AR agonists decrease keratinocytes' ability to respond, further implicating the use of topical timolol for recalcitrant wounds. Angiogenesis and dermal fibroblast proliferation are also regulated by B2ARs. The B2AR antagonists have been found to promote angiogenesis in chick chorioallantoic membrane assays and in vivo murine wound models. Dermal fibroblast migration is also increased (by 27%) when exposed to B2AR antagonists, and epidermal differentiation is improved with B2AR antagonists and β1- and β2-receptor antagonists.

Full-thickness skin grafts (FTSG) are one of the most commonly performed procedures in dermatologic, plastic and burn surgery. Various experimental approaches to optimize the healing of FTSG receiving sites have been described; however, no clearly superior and easily applicable method has gained wide acceptance in daily practice.

As indicated by preliminary evidence in other wound healing endeavors, 0.25% timolol gel may represent a commercially available, safe and simple, painless and relatively inexpensive treatment for improving healing of FTSG receiving site, as well as for improving cosmetic long term outcomes.

To assess the efficacy and safety of topically applied 0.25% timolol gel in promoting wound healing in FTSG receiving site versus standard of care (SOC) by:

1. Evaluating healing in response to treatment with 0.25% topical timolol gel versus SOC in terms of wound surface area and Graft Take Score at the receiving site of a FTSG at 7 and 14 days;
2. Evaluating cosmetic outcomes of the receiving site of a FTSG in terms of blinded physician (Vancouver Scar Scale, VSS) and patient (Visual Analogue Scale, VAS) assessment at 3 and 6 months' follow up;
3. Evaluating the need for further scar revision (dermabrasion or pulsed dye laser [PDL]) at the 6-month follow up;
4. Evaluating patient discomfort during the healing process by means of a patient pain VAS; and
5. Determining the side effects associated with 0.25% timolol gel versus SOC

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Undergoing a procedure which results in the need of a FTSG
3. Willing to provide written informed consent

Exclusion Criteria:

1. Age less than 18 years of age
2. Pregnant women
3. (Use of systemic drugs that can impede wound healing, such retinoids or immune-suppressive drugs)
4. Severe coagulation disorders
5. Severe, uncontrolled systemic comorbidities, such as diabetes, arthritis, etc.
6. Hypersensitivity to 0.25% timolol gel
7. Not willing to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Evaluating the need for further scar revision (via dermabrasion or pulsed dye laser (PDL)) | 6-months' post-surgery
  A study physician will review the healed scar site to determine if there are potential cosmetic factors that could be improved through scar revision. If the patient is interested in having scar revision procedures, the study physician will offer a dermabrasion or PDL to treat the scar site.

SECONDARY OUTCOMES:
Evaluating cosmetic outcomes of the receiving site of a FTSG via Vancouver Scar Scale (VSS) | 3 months' post-surgery and 6 months' post-surgery
  Physician blinded to subject's treatment group uses VSS which documents scar appearance change over time via photos. VSS ranges from 0 (most desirable outcome) to 13 (least desirable). A lower score is considered a better outcome and a higher score is a worse outcome. VSS consists of 4 sub-scales, with each reporting a value. The "pigmentation" ranges from 0 (normal pigment) to 2 (hyperpigment); "vascularity" ranges from 0 (normal appearance) to 3 (purple appearance); "pliability" ranges from 0 (normal) to 5 (contracture); "height" ranges from 0 (normal/flat) to 3 (>5mm). Sub-scale scores are combined to give an overall VSS score.
Evaluating cosmetic outcomes of the receiving site of a FTSG via patient Visual Analogue Scale (VAS) | 3 months' post-surgery and 6 months' post-surgery
  Scar VAS rates subjects' graft cosmetic appearance. Each question ranges from 1 (no complaints w/ itch or pain/as normal skin) to 10 (worst imaginable itch or pain/very different from normal skin). Ranges from 6 (best outcome score) to 66 (worst outcome score); a lower score is considered a better outcome and a higher score is considered a worse outcome.
Evaluating change in healing response to treatment with 0.25% topical timolol gel versus SOC in terms of wound surface area at the receiving site of a FTSG via Graft Take Score | 7 days post-surgery, and 14 days post-surgery
  The Graft Take Score will be used to assess amount of graft take at each visit. Graft take is considered "Good" if 90%+ of the graft site is healed and pink/purple in color; "Moderate" if there is 50% healing, pink or purple in color, and >50% of the graft has taken; and "Poor" if <50% graft take.
Evaluating change in healing response to treatment with 0.25% topical timolol gel versus SOC in terms of wound surface area at the receiving site of a FTSG via histogram planimetry | 7 days post-surgery, and 14 days post-surgery
  Histogram planimetry is more accessible than automated analysis software programs, and it is based on the pixel count of a selected irregular area which is divided by the pixel count of 1 cm2 to find a result in terms of cm2 or mm2.
Evaluating change in patient discomfort during the healing process by means of a patient pain VAS | 7 days' post-surgery, 14 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery
  Subjects will be asked to complete a Visual Analogue Scale for scar assessment to rate how they think their graft sites appear cosmetically compared to normal skin, and any complaints about how painful they sites are, and how itchy they feel. Each question ranges from 1 (no complaints with itch or pain/as normal skin) to 10 (worst imaginable itch or pain/very different from normal skin). The score ranges from 6 (best outcome score) to 66 (worst outcome score), thus a lower score is considered to have a better outcome and a higher score is considered a worse outcome.
Determining change in the side effects associated with 0.25% timolol gel versus SOC via physician assessment | 7 days' post-surgery, 14 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery
  A physician will assess for side effects and determine whether they are likely associated with the 0.25% topical timolol or part of the normal wound healing experience.
Determining change in the side effects associated with 0.25% timolol gel versus SOC via patient assessment | 7 days' post-surgery, 14 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery
  Patients will report any side effects they experience post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mohs and Dermatologic Surgery Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided